CLINICAL TRIAL: NCT01519856
Title: Efficacy and Safety of Long-term Therapy With Piribedil (CLARIUM) in Patients With M. Parkinson Under Consideration of Quality of Life Parameters and Cognitive Function
Brief Title: PIRLONG-PD Safety and Efficacy of Piribedil in Parkinson's Disease During Long Term Therapy
Acronym: PIR-008/K
Status: Completed | Type: Observational
Sponsor: Desitin Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PIR-008/K
Record Dates: First submitted 2010-03-12; First posted 2012-01-27 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson's Disease
Keywords: open; non-intervention; observational
MeSH Terms: conditions — Parkinson Disease | interventions — Piribedil; Loratadine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tablet
  Interventions: Drug: piribedil (Clarium)

INTERVENTIONS:
Drug: piribedil (Clarium) — oral tablets, 50 mg

SUMMARY:
Non-Ergot Dopamine agonists are meanwhile the drugs of first-choice in the treatment of Parkinson's disease. The receptor profile of the non-ergot dopamine-agonist piribedil is unique. In addition to agonistic effects on dopaminergic D2- and D3-receptors piribedil has adrenergic alpha-2A- and alpha-2C-receptors antagonisic properties. There is evidence from the literature that the antagonistic properties of piribedil are correlated with an improvement of cognitive function and vigilance parameters in parkinson's disease. The aim of the present non-interventional study is to investigate the safety and efficacy of piribedil during long-term therapy of patients with M. Parkinson under consideration of cognitive functions and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed or advanced idiopathic Parkinson's disease
* male and female patients over 18 years of age
* indication for treatment with piribedil according to Summary of Product Characteristics (SmPC)

Exclusion Criteria:

* in line with piribedil SmPC
* in particular hypersensitivity to piribedil or to any of the excipients and pregnancy and lactation as stated in the SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female patients with Morbus Parkinson
Sampling Method: Non-Probability Sample
Enrollment: 908 (Actual)
Dates: Start 2009-06; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Adverse event profile during long term therapy with piribedil in patients with Parkinson's disease | 4 years

SECONDARY OUTCOMES:
Influence on quality of life | 4 years
Quality of life parameters | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Erich Scholz, Böblingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Castro-Caldas A, Delwaide P, Jost W, Merello M, Williams A, Lamberti P, Aguilar M, Del Signore S, Cesaro P; Parkinson-Control Study Group. The Parkinson-Control study: a 1-year randomized, double-blind trial comparing piribedil (150 mg/day) with bromocriptine (25 mg/day) in early combination with levodopa in Parkinson's disease. Mov Disord. 2006 Apr;21(4):500-9. doi: 10.1002/mds.20750. PMID 16267842
- [Background] Rascol O, Dubois B, Caldas AC, Senn S, Del Signore S, Lees A; Parkinson REGAIN Study Group. Early piribedil monotherapy of Parkinson's disease: A planned seven-month report of the REGAIN study. Mov Disord. 2006 Dec;21(12):2110-5. doi: 10.1002/mds.21122. PMID 17013922
- [Background] Peretti CS, Gierski F, Harrois S. Cognitive skill learning in healthy older adults after 2 months of double-blind treatment with piribedil. Psychopharmacology (Berl). 2004 Nov;176(2):175-81. doi: 10.1007/s00213-004-1869-8. Epub 2004 May 12. PMID 15138753
- [Background] Schuck S, Bentue-Ferrer D, Kleinermans D, Reymann JM, Polard E, Gandon JM, Allain H. Psychomotor and cognitive effects of piribedil, a dopamine agonist, in young healthy volunteers. Fundam Clin Pharmacol. 2002 Feb;16(1):57-65. doi: 10.1046/j.1472-8206.2002.00070.x. PMID 11903513